CLINICAL TRIAL: NCT00382200
Title: Phase I/II Study of Decitabine and All-Trans Retinoic Acid (Tretinoin) for Patients With Myelodysplastic Syndromes
Brief Title: Decitabine and Tretinoin in Treating Patients With Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-054; MSKCC-06054
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Results first posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2023-01

CONDITIONS: Myelodysplastic Syndromes
Keywords: de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Decitabine; Tretinoin; DNA Methylation; Cytogenetic Analysis; Microarray Analysis; Flow Cytometry; Immunohistochemistry

ARMS (1):
- Decitabine and All-Trans Retonoic Acid (Tretinoin) (Experimental): Decitabine and All-Trans Retonoic Acid (Tretinoin)
  Interventions: Drug: decitabine; Drug: tretinoin; Genetic: DNA methylation analysis; Genetic: cytogenetic analysis; Genetic: microarray analysis; Other: flow cytometry; Other: immunohistochemistry staining method

INTERVENTIONS:
Drug: decitabine
Drug: tretinoin
Genetic: DNA methylation analysis
Genetic: cytogenetic analysis
Genetic: microarray analysis
Other: flow cytometry
Other: immunohistochemistry staining method

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as decitabine, work in different ways to stop the growth of myelodysplastic cells, either by killing the cells or by stopping them from dividing. Tretinoin and decitabine may help myelodysplastic cells become more like normal cells, and to grow and spread more slowly. Giving decitabine together with tretinoin may be an effective treatment for myelodysplastic syndromes.

PURPOSE: This phase I/II trial is studying the side effects and best dose of tretinoin when given together with decitabine in treating patients with myelodysplastic syndromes.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the hematologic and nonhematologic toxicities of decitabine in combination with tretinoin in patients with myelodysplastic syndromes. (Phase I)
* Determine the maximum tolerated dose of tretinoin when administered with decitabine in these patients. (Phase I)
* Determine the clinical remission rate (complete and partial remission) in patients treated with this regimen. (Phase II)
* Determine the rate of hematologic improvement in these patients. (Phase II)

Secondary

* Determine the efficacy of this regimen, in terms of improved bone marrow function, by monitoring frequency of transfusion, bleeding, and infection, as well as changes in bone marrow morphology and cytogenetics in these patients.
* Assess differentiation by morphology and flow cytometry and apoptosis by flow cytometry in patients treated with this regimen.
* Determine if gene expression changes in these patients are induced by this regimen.
* Determine the efficacy of this regimen, in terms of inducing demethylation of specific genes, in these patients.
* Correlate clinical response with gene expression, demethylation of specific genes, and flow cytometric indicators of differentiation and apoptosis.

OUTLINE: This is a phase I, dose-escalation study of tretinoin followed by a phase II, open-label study.

* Phase I: Patients receive decitabine IV over 1 hour once daily on days 1-5 followed by oral tretinoin twice daily on days 10-19. Treatment repeats every 28 days for a minimum of 4 courses in the absence of disease progression or excessive toxicity. Patients who achieve a partial or complete response after completing 6 courses of treatment may receive 4 additional courses up to a total of 10 courses. Patients with stable disease or hematologic improvement are removed from study.

Cohorts of 3-6 patients receive escalating doses of tretinoin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity attributable to tretinoin at any dose level during course 1. A total of 6 patients are treated at the MTD.

* Phase II: Patients receive decitabine as in phase I and tretinoin at the MTD. Patients undergo blood and bone marrow collection periodically during study for correlative demethylation and gene profiling studies and for evidence of differentiation and apoptosis. Samples are examined by flow cytometry, cytogenetics, histochemistry, and array-based whole genome methylation analysis.

After completion of study treatment, patients are followed at 30 days.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed myelodysplastic syndromes (MDS)
* International Prognostic scoring system (IPSS) score ≥ 0.5, including the following:

  * Untreated or treated intermediate-1 risk disease
  * Intermediate-2 risk disease
  * High-risk disease
* No treatment-related MDS
* Ineligible for transplantation
* No decitabine-refractory disease defined as disease progression after discontinuation of therapy

  * If previously treated with decitabine, must have responded to therapy (hematologic improvement or better per International Working Group Response Criteria)

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Bilirubin ≤ 2.5 mg/dL
* AST and ALT ≤ 2 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other medical condition that, in the opinion of the treating physician, would preclude patient compliance or put patient at excessive risk of treatment-related toxicity
* No other malignancy that would likely require systemic chemotherapy within 4 months after starting study treatment
* No allergy to parabens, vitamin A, or retinoids

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior azacytidine allowed
* More than 4 weeks since prior cytotoxic chemotherapy or radiotherapy
* More than 4 weeks since prior experimental therapy
* Concurrent myeloid growth factors allowed only in the setting of febrile neutropenia according to established guidelines for use

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-07; Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raajit Rampal, MD, PhD, Study Chair — Memorial SloanKettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Tretinoin 45 mg/m2/Day; Phase I: Tretinoin 65 mg/m2/Day; Phase I: Tretinoin 85 mg/m2/Day; Phase II: MTD Tretinoin 65 mg/m2/Day: Decitabine and All-Trans Retonoic Acid (Tretinoin)
Period: Overall Study
Arm/Group | Phase I: Tretinoin 45 mg/m2/Day | Phase I: Tretinoin 65 mg/m2/Day | Phase I: Tretinoin 85 mg/m2/Day | Phase II: MTD Tretinoin 65 mg/m2/Day
Started | 5 | 14 | 7 | 28
Completed | 5 | 14 | 7 | 28
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decitabine and All-Trans Retonoic Acid (Tretinoin) | Phase I: Tretinoin 65 mg/m2/Day | Phase I: Tretinoin 85 mg/m2/Day | Phase II: MTD Tretinoin 65 mg/m2/Day | Total
Number analyzed (Participants) | 5 | 14 | 7 | 28 | 54
Age, Continuous [Median (Full Range); unit: years] | 71 [52 to 72] | 66.5 [44 to 77] | 64 [33 to 78] | 66.5 [45 to 83] | 68 [33 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 8 | 15
  Male | 3 | 12 | 4 | 20 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 0 | 3
  Not Hispanic or Latino | 3 | 14 | 6 | 28 | 51
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 5 | 11 | 7 | 28 | 51
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 14 | 7 | 28 | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Evaluated for Hematologic and Nonhematologic Toxicities as Measured by NCI CTC v2.0
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Tretinoin 45 mg/m2/Day | Phase I: Tretinoin 65 mg/m2/Day | Phase I: Tretinoin 85 mg/m2/Day | Phase II: MTD Tretinoin 65 mg/m2/Day
Number analyzed (Participants) | 5 | 14 | 7 | 28
Participants | 5 | 14 | 7 | 28

2. Primary Outcome: Maximum Tolerated Dose of Tretinoin When Administered With Decitabine as Determined by NCI CTC v2.0 (Phase II)
Time Frame: Up to 1 year
Measure: Number; unit: mg/m^2/day of tretinoin
Arm/Group | Phase II: MTD Tretinoin 65 mg/m2/Day
Number analyzed (Participants) | 28
mg/m^2/day of tretinoin | 65

3. Primary Outcome: Overall Response Rate
Description: Overall Response Rate is defined as Complete Response + Partial Response
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Tretinoin 45 mg/m2/Day | Phase I: Tretinoin 65 mg/m2/Day | Phase I: Tretinoin 85 mg/m2/Day | Phase II: MTD Tretinoin 65 mg/m2/Day
Number analyzed (Participants) | 5 | 14 | 7 | 28
Participants
  Participants with either Complete or Partial Response | 4 | 6 | 2 | 13
  Participants Evaluated without Complete or Partial Response | 0 | 4 | 1 | 11
  Not Evaluable for Response | 1 | 4 | 4 | 4

4. Primary Outcome: Rate of Hematologic Improvement as Measured by Responding Cell Lines (Erythroid, Platelet, and Neutrophil Response) (Phase II)
Time Frame: After each cycle
Population: N/A data were not collected
Arm/Group | Decitabine and All-Trans Retonoic Acid (Tretinoin)
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Bone Marrow Function as Measured by Frequency of Transfusion, Bleeding, and Infection as Well as Changes in Bone Marrow Morphology and Cytogenetics
Time Frame: After each cycle
Population: N/A data were not collected
Arm/Group | Decitabine and All-Trans Retonoic Acid (Tretinoin)
Number analyzed (Participants) | 0

6. Secondary Outcome: Differentiation as Measured by Morphology and Flow Cytometry and Apoptosis as Measured by Flow Cytometry
Time Frame: After each cycle
Population: N/A data were not collected
Arm/Group | Decitabine and All-Trans Retonoic Acid (Tretinoin)
Number analyzed (Participants) | 0

7. Secondary Outcome: Gene Expression Changes as Measured by Affymetrix Gene Profiling Studies
Time Frame: After each cycle
Population: N/A data were not collected
Arm/Group | Decitabine and All-Trans Retonoic Acid (Tretinoin)
Number analyzed (Participants) | 0

8. Secondary Outcome: Demethylation of Specific Genes as Measured by Gene Promoter Methylation Studies
Time Frame: After each cycle
Population: N/A data were not collected
Arm/Group | Decitabine and All-Trans Retonoic Acid (Tretinoin)
Number analyzed (Participants) | 0

9. Secondary Outcome: Correlation of Clinical Response, With Gene Expression, Demethylation of Specific Genes, and Flow Cytometric Indicators of Differentiation and Apoptosis
Time Frame: After each cycle
Population: N/A data were not collected
Arm/Group | Decitabine and All-Trans Retonoic Acid (Tretinoin)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 1 year
Arm/Group | Phase I: Tretinoin 45 mg/m2/Day | Phase I: Tretinoin 65 mg/m2/Day | Phase I: Tretinoin 85 mg/m2/Day | Phase II: MTD Tretinoin 65 mg/m2/Day
All-Cause Mortality (participants affected / at risk) | 0/5 | 2/14 | 1/7 | 10/28
Serious Adverse Events (participants affected / at risk) | 5/5 | 9/14 | 5/7 | 21/28
Other Adverse Events (participants affected / at risk) | 5/5 | 14/14 | 7/7 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Tretinoin 45 mg/m2/Day (N=5) | Phase I: Tretinoin 65 mg/m2/Day (N=14) | Phase I: Tretinoin 85 mg/m2/Day (N=7) | Phase II: MTD Tretinoin 65 mg/m2/Day (N=28)
Abdominal pain/cramping (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Bilirubin (Investigations) | 0 | 0 | 1 | 0
Blood, bone marrow, other (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Cardiovascular, Arrhythmia, other (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiovascular, other (Cardiac disorders) | 0 | 0 | 0 | 2
Chest pain (Cardiac disorders) | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Creatinine (Investigations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Derm, skin other (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Dyspnea (Reproductive system and breast disorders) | 1 | 1 | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0
Edema (General disorders) | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 6 | 3 | 10
Fever (General disorders) | 0 | 0 | 0 | 1
Gastrointestinal, other (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Infection without neutropenia (Infections and infestations) | 0 | 1 | 0 | 2
Infection with febrile neutropenia (Blood and lymphatic system disorders) | 2 | 3 | 2 | 8
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Neutrophils (Investigations) | 0 | 0 | 1 | 2
Pain (General disorders) | 1 | 0 | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 2
Typhlitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0
Wound, infectious (Infections and infestations) | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 2 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Tretinoin 45 mg/m2/Day (N=5) | Phase I: Tretinoin 65 mg/m2/Day (N=14) | Phase I: Tretinoin 85 mg/m2/Day (N=7) | Phase II: MTD Tretinoin 65 mg/m2/Day (N=28)
Platelets (Investigations) | 3 | 7 | 4 | 28
Neutrophils (Investigations) | 4 | 11 | 6 | 24
Hemoglobin (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 11
Leukocytes (Investigations) | 5 | 13 | 7 | 28
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 4 | 0 | 12
ALT (Investigations) | 0 | 3 | 0 | 3
Headache (Nervous system disorders) | 0 | 1 | 2 | 0
AST (Investigations) | 0 | 1 | 1 | 4
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 | 5 | 3 | 9
Alkaline Phosphatase (Investigations) | 0 | 0 | 1 | 1
Lymphopenia (Investigations) | 2 | 11 | 6 | 22
Bilirubin (Investigations) | 1 | 1 | 2 | 5
Rash, desquamation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Creatinine (Investigations) | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Infection with grade 3/4 neutr (Infections and infestations) | 3 | 4 | 2 | 4
Derm, skin other (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 10
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 5 | 2 | 10
Infection w/out neutropenia (Infections and infestations) | 0 | 0 | 0 | 4
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 1 | 0 | 0
Fever (General disorders) | 0 | 0 | 0 | 0
Hypermagnemesia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 3
PTT (Investigations) | 0 | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 1 | 0
PT (Investigations) | 0 | 0 | 0 | 5
Amylase (Investigations) | 1 | 0 | 0 | 0
Lipase (Investigations) | 1 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Blood bicarbonate (Investigations) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 4 | 0 | 0
Hypotention (Vascular disorders) | 0 | 2 | 0 | 0
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Typhlitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
GI, other (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Fibrinogen (Investigations) | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hypernatremia (Investigations) | 0 | 0 | 0 | 1
Hypoglycemia (Investigations) | 0 | 0 | 0 | 1
Pulmonary, other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT00382200/Prot_SAP_000.pdf